CLINICAL TRIAL: NCT03502473
Title: Clinical Assessment to Evaluate UltraShape Power Device Performance for Flanks Fat Reduction
Brief Title: UltraShape Power Device for Fat Reduction in Flanks
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision was made not to initiate and to focus on other initiatives
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHF24961
Record Dates: First submitted 2018-03-20; First posted 2018-04-18 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Excess Abdominal Fat
Keywords: fat flanks

STUDY DESIGN:
Intervention Model Description: Flanks will be randomized in accordance with randomization list. One flank will receive a single treatment pass or no treatment. The other side will receive multiple passes (up to 5 passes) during the same treatment session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- One pass/no treatment arm (Experimental): One random flank will be treated with UltraShape Power device with one pass or remained as a control (no treatment)
  Interventions: Device: UltraShape Power device
- Multiple passes treatment arm (Experimental): Second flank will be treated with UltraShape Power device with multiple passes.
  Interventions: Device: UltraShape Power device

INTERVENTIONS:
Device: UltraShape Power device — UltraShape Power is a non-invasive focused ultrasound device, approved by the FDA (160896K;170370K); CE; Israeli Ministry of Health. The UltraShape Power system works by emitting acoustic waves of focused ultrasonic energy (200 ± 30 KHz frequency) that converge into a confined focal volume underneath the skin, thereby, targeting only subcutaneous fat at a controlled depth. Unlike traditional ultrasound technology, UltraShape Power's energy transmits pulsed ultrasound, allowing control over temperature elevation. The system comprised of two main parts:
  * The Main console
  * Transducer

SUMMARY:
Prospective, baseline-controlled evaluation of the UltraShape Power device for non-invasive fat reduction in flanks.

DETAILED DESCRIPTION:
Eligible subjects will receive 3 bi-weekly treatments (2 weeks interval) with the UltraShape Power device according to the study protocol.

One random flank will be treated with one pass or remained as a control (no treatment) while the second flank will be treated with multiple passes.

Subjects will return for up to 4 follow up visits: 4 weeks, 8 weeks, 12 weeks and (optional) 24 weeks following end of treatment/s.

Each subject will be enrolled for total expected study duration of up to 28 weeks.

After last follow up visit, subjects who wish will receive compensation treatments (up to 3) on the flank who received regular treatment (single pass) or remained as a control (no treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Female and male subjects, 18 and 65 years of age at the time of enrolment
3. Fitzpatrick Skin Type I to VI.
4. Fat thickness of at least 1.5 cm in the treated area (measured by calibrated caliper).
5. BMI interval: 19 ≤ BMI ≤ 30 (normal to overweight, but not obese).
6. If female, not pregnant, lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
7. In addition, negative pregnancy inquiry as reviewed before each treatment and each follow up visit for women with bearing potential (e.g. not menopause).
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
10. Willingness to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
11. Willing to have photographs and images taken of the treated areas to be used de-identified in evaluations, publications and presentations.

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism
2. Current hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions
4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone
6. Having undergone any other surgery in the treated areas within 3 months of treatment or during the study, including liposuction
7. Previous body contouring procedures in the treatment area within 12 months
8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
9. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
10. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
11. Very poor skin quality (i.e., severe laxity)
12. Abdominal wall diastasis or hernia on physical examination
13. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
14. Obesity (BMI > 30)
15. Childbirth within the last 12 months or breastfeeding women. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
16. Unstable weight within the last 6 months (i.e., ± 3% weight change in the prior six months)
17. Inability to comply with fat measurement procedures (e.g., inability to hold breath for few seconds).
18. Fat thickness lower than 1.5 cm before strapping at the treated area.
19. Participation in another clinical study involving same anatomical areas within the last 6 months (or 30 days in case different anatomical areas were treated in previous trial/s).
20. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-03-07 (Estimated); Study Completion 2019-09-07 (Estimated)

PRIMARY OUTCOMES:
Fat Volume reduction | 12 weeks follow-up (12wk FU) versus baseline
  MRI measurements for fat thickness in cc (cubic centimeter)
Treatment Safety as Assessed by Blood Lipid Level | up to 24 weeks
  Verification similar of post-treatment and pre-treatment (baseline) blood lipid levels values [%]

SECONDARY OUTCOMES:
MRI Measurement of Fat Thickness Reduction | 4 weeks, 8 weeks, 12 weeks and (optional) 24 weeks versus baseline.
  MRI measurements for Fat thickness in mm
Ultrasound Measurement of Fat Thickness Reduction | 4 weeks, 8 weeks, 12 weeks and (optional) 24 weeks versus baseline.
  Ultrasound measurements for Fat thickness in mm
Fat Volume reduction | 4 weeks, 8 weeks and (optional) 24 weeks versus baseline.
  MRI measurements for fat thickness in cc (cubic centimeter)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jerdev, MD, Principal Investigator — The Baruch Padeh Medical Center
Locations (1):
- The Baruch Padeh Medical Center, Tiberias, Israel

IPD SHARING:
Plan to Share IPD: No